CLINICAL TRIAL: NCT01344525
Title: Pilot Project on Interdisciplinary Therapy of Obesity and Its Consequences on Body Weight, Quality of Life and Gastrointestinal Parameters
Brief Title: Pilot Project on Interdisciplinary Therapy of Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: OGIT-FKZ01GI0843
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Obesity; Weight Loss
Keywords: obesity therapy; metabolic syndrome; gastrointestinal tract; microbiota; metabolomics; micronutrients; outcome; sustainability
MeSH Terms: conditions — Obesity; Weight Loss; Metabolic Syndrome | interventions — Anastomosis, Roux-en-Y

ARMS (4):
- Control group (No Intervention): Nutritional counselings every 6 months, no further intervention
- "low-calorie-diet (LCD)"-based lifestyle intervention (Experimental): 12 months multidisciplinary weight loss program including three months low-calorie formula diet (800 kcal) (OPTIFAST®52 program)
  Interventions: Procedure: Multidisciplinary lifstyle intervention
- Laparoscopic gastric sleeve intervention (Experimental)
  Interventions: Procedure: Laparoscopic gastric sleeve
- Conventional bariatric surgery (Experimental): Gastric Banding and Gastric Bypass
  Interventions: Procedure: Gastric Banding; Procedure: Roux-en-Y Bypass

INTERVENTIONS:
Procedure: Laparoscopic gastric sleeve — Laparoscopic gastric sleeve
  Arms: Laparoscopic gastric sleeve intervention
Procedure: Gastric Banding — Gastric Banding
  Arms: Conventional bariatric surgery
Procedure: Multidisciplinary lifstyle intervention — Multidisciplinary lifstyle intervention (OPTIFAST®52-program)
  Arms: "low-calorie-diet (LCD)"-based lifestyle intervention
Procedure: Roux-en-Y Bypass — Roux-en-Y Bypass
  Arms: Conventional bariatric surgery

SUMMARY:
Obese individuals that undergo major intervention such as a low-calorie formula diet program or bariatric surgery with the result of substantial weight loss (> 10%) are included and followed-up for at least 3 years. Weight changes and excess weight loss as well as measures of quality of life are monitored. In addition, biomaterials will be collected from these individuals every 6 months for measurement of parameters related to obesity-associated gastrointestinal (GI) impairments such as change in GI hormone levels, change in GI microbiota, or enhanced bacterial translocation. Moreover, micronutrient and metabolomics analysis will be performed. This project allows comparison of non-surgical and surgical intervention and enables to asses the anticipated relationship between obesity and the GI tract in humans in the future.

DETAILED DESCRIPTION:
A database and a biomaterial bank will be established to assess, if the role of the gut for the development of obesity and obesity-related diseases such as fatty liver are of relevance in humans, e.g. for classification of afflicted individuals regarding risk or outcome after intervention. During 3 years, the investigators will include 480 obese individuals (4 cohorts of 120 individuals) who undergo a treatment program (either surgical or non-surgical), and follow them up for at least 3 years. Every 6 months, a visit is planned at the obesity center where the initial intervention has been performed. Within the visits, anthropometry (Body Mass Index (BMI), excess body weight (EBW), bioelectrical impedance analysis (BIA)), quality of life (SF36 score, Impact Of Weight On Quality Of Life (IWQOL) questionnaire), and sample collection for laboratory analyses (inflammatory markers, hormones, flora composition, micronutrients, metabolomics etc.) will be performed. Patients will be recruited from 3 centers in Germany. The long-term expectation from this model project is to find gastrointestinal parameters allowing to predict outcome and sustainability of different intervention strategies. In addition, intervention programs will be compared regarding long-term outcome and quality of life changes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-65 years at time of inclusion)
* Obesity defined as BMI > 30 kg/m2
* Obesity treatment (multidisciplinary life style intervention with LCD or bariatric surgery) resulting in an estimated body weight loss of >10% of the initial body weight within 6 month

Exclusion Criteria:

* Body weight loss after intervention < 10%
* Follow-up period < 1 year or number of consultations within 3 years < 3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2009-05; Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Body weight loss | Every 6 months for a period of 3 years

SECONDARY OUTCOMES:
Quality of life | Every 6 months for a period of 3 years
  SF-36, IWQOL-lite
Physical examination | Every 6 months for a period of 3 years
  Weight, height, waist circumference, blood pressure, bioelectric impedance analysis, pulse etc.
Laboratory analysis | Every 6 months for a period of 3 years
  Fasting glucose; Glutamat-Pyruvat- Transaminase (GPT); Lipid parameters (cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, triglycerides)
Vitamins/micronutrients | Every 3-6 months for a period of maximal 3 years
  Vitamin B1, B6, B12, ß-carotene, niacin, folic acid, selen and oxidative metabolites
Metabolomics, and Microflora analysis | Every 3-6 months for a period of maximal 3 years
Liver fat | Every 6 months for a period of 3 years
  Liver sonography
gut permeability | Every 6 months for a period of 3 years
  assessed by the uptake of inert molecules
peripheral blood lipopolysaccharide concentrations | Every 6 months for a period of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C. Bischoff, Prof. Dr., Principal Investigator — University of Hohenheim, Institute of Nutritional Medicine
Locations (3):
- Germany (3):
  - University of Heidelberg, Heidelberg
  - University of Hohenheim, Stuttgart
  - University of Tübingen, Tübingen

REFERENCES:
- [Derived] Damms-Machado A, Louis S, Schnitzer A, Volynets V, Rings A, Basrai M, Bischoff SC. Gut permeability is related to body weight, fatty liver disease, and insulin resistance in obese individuals undergoing weight reduction. Am J Clin Nutr. 2017 Jan;105(1):127-135. doi: 10.3945/ajcn.116.131110. Epub 2016 Nov 9. PMID 28049662
- [Derived] Damms-Machado A, Mitra S, Schollenberger AE, Kramer KM, Meile T, Konigsrainer A, Huson DH, Bischoff SC. Effects of surgical and dietary weight loss therapy for obesity on gut microbiota composition and nutrient absorption. Biomed Res Int. 2015;2015:806248. doi: 10.1155/2015/806248. Epub 2015 Feb 1. PMID 25710027
- [Derived] Damms-Machado A, Weser G, Bischoff SC. Micronutrient deficiency in obese subjects undergoing low calorie diet. Nutr J. 2012 Jun 1;11:34. doi: 10.1186/1475-2891-11-34. PMID 22657586
- [Derived] Damms-Machado A, Friedrich A, Kramer KM, Stingel K, Meile T, Kuper MA, Konigsrainer A, Bischoff SC. Pre- and postoperative nutritional deficiencies in obese patients undergoing laparoscopic sleeve gastrectomy. Obes Surg. 2012 Jun;22(6):881-9. doi: 10.1007/s11695-012-0609-0. PMID 22403000